CLINICAL TRIAL: NCT03301857
Title: Long-term Safety Follow-up of Subjects With Giant Cell Tumor of Bone Treated With Denosumab in Study 20062004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20140114; 2017-001758-32 (EudraCT Number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Participants who are still being treated with denosumab when 20062004 completes: 120 mg administered subcutaneously (SC) every 4 weeks (Q4W).
  For participants undergoing retreatment with denosumab: 120 mg administered SC on Days 1, 8, 15 and 28 then every 4 weeks subsequently.
  Interventions: Drug: Denosumab
- Safety Follow-up (No Intervention): Participants who completed denosumab treatment and were in safety follow-up at the conclusion of 20062004 will have follow-up visits performed every 6 months via telephone or in-person clinic visit.

INTERVENTIONS:
Drug: Denosumab — 120 mg administered subcutaneously (SC) every 4 weeks (Q4W).
  Other Names: AMG 162, Immunoglobulin G2 human monoclonal antibody to RANK ligand
  Arms: Denosumab

SUMMARY:
Study 20140114 will continue to follow participants with GCTB who were treated in Study 20062004 and remained on the study at the completion of Study 20062004 for an additional 5 years on long-term safety follow up.

DETAILED DESCRIPTION:
Study 20140114 will continue to follow participants with GCTB who were treated in Study 20062004 and remained on the study at the completion of Study 20062004 for an additional 5 years on long-term safety follow up. Collection of long-term safety information will include adverse events of interest and all treatment-emergent adverse events and serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Participant was previously enrolled in Study 20062004.
* Participant or participant's legally acceptable representative has provided informed consent/assent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* Females of childbearing potential on denosumab and not willing to continue to use 1 highly effective method of contraception during treatment and for 5 months after the end of treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (5):
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - Washington Cancer Institute at MedStar Washington Hospital, Washington D.C., District of Columbia
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mount Sinai Beth Israel Downtown, New York, New York
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Istituti Ortopedici Rizzoli, Bologna, Italy
- Poland (2):
  - Instytut Matki i Dziecka, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie â€" Panstwowy Instytut Badawczy, Warsaw
- Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands, Spain
- Skane Universitetssjukhus, Lund, Sweden
- Royal Orthopaedic Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with giant cell tumor of bone (GCTB) were enrolled across 8 countries (Australia, Italy, France, Poland, Spain, Sweden, the United Kingdom of Great Britain and Northern Ireland, and the United States) between November 2017 and July 2023.
Pre-assignment Details: Participants in the study were enrolled upon completing study 20062004.
Groups:
- Exposed to Investigational Product (IP): Participants who received denosumab at the conclusion of study 20062004 continued in this study (study 20140114), and received denosumab at the current dose (120 mg every 4 weeks [Q4W] subcutaneous injection [SC]) and schedule at the investigator's discretion.
- Not Exposed to IP: Participants who completed denosumab treatment in study 20062004 and were in the safety follow up at the conclusion of study 20062004 continued in long term safety follow up in this study (study 20140114), and did not receive denosumab.
Period: Overall Study
Arm/Group | Exposed to Investigational Product (IP) | Not Exposed to IP
Started | 51 | 34
Received Denosumab | 51 | 0
Completed | 29 | 26
Not Completed | 22 | 8
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Decision by Sponsor | 6 | 0
Not completed — Withdrawal by Subject | 12 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants (from study 20062004) who provided informed consent and had a non-missing enrolment date in this study.
Groups:
- Exposed to IP: Participants who received denosumab at the conclusion of study 20062004 continued in this study (study 20140114), and received denosumab at the current dose (120 mg Q4W SC) and schedule at the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Exposed to IP | Not Exposed to IP | Total
Number analyzed (Participants) | 51 | 34 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (12.8) | 46.7 (15.1) | 44.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 23 | 55
  Male | 19 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 38 | 24 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 31 | 66
  Other | 10 | 0 | 10
  Black (or African American) | 4 | 3 | 7
  Asian | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) of Interest (EOI)
Description: EOIs assessed in the study were signs and symptoms of osteonecrosis of the jaw (ONJ), malignancy (including malignancy in GCTB), atypical femoral fracture (AFF), hypocalcemia, hypercalcemia after treatment discontinuation, pregnancy and lactation (if occurring during treatment or within 5 months of the last dose of denosumab). Hypocalcemia includes events that occurred after 30 days following the last dose of IP and includes TEAEs only. Other EOIs encompass all events from signing the informed consent to the end of the study (approximately 5 years). ONJ and AFF events were adjudicated by independent reviewers.
Time Frame: Up to approximately 5 years
Population: FAS included all enrolled participants (from study 20062004) who provided informed consent and had a non-missing enrolment date in this study.
Measure: Number; unit: Count of Participants
Arm/Group | Exposed to IP | Not Exposed to IP
Number analyzed (Participants) | 51 | 34
Count of Participants
  Adjudicated positive ONJ | 3 | 0
  Malignancy, including malignancy in GCTB | 6 | 1
  Adjudicated positive AFF | 2 | 0
  Hypocalcemia | 3 | 0
  Hypocalcemia after treatment end | 0 | 0
  Pregnancy and lactation | 0 | 0

2. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAE)
Description: An AE is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. An AE is considered as treatment-emergent if the AE occurs during the time period from the first dose of IP in this study through last dose of IP plus 30 days. TEAEs related to IP include only TEAEs for which the Investigator indicated there was a reasonable possibility they may have been caused by IP. AEs were graded (grade 3 [severe or medically significant but not immediately life-threatening], 4 [life-threatening], and 5 [death related to the AE]) using the Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Measure: Number; unit: Count of Participants
Arm/Group | Exposed to IP
Number analyzed (Participants) | 51
Count of Participants
  All TEAEs | 47
  Serious TEAEs | 8
  Fatal TEAEs | 0
  TEAEs leading to IP discontinuation | 9
  CTCAE Grade 3, 4, or 5 | 16
  All TEAEs related to IP | 14

3. Secondary Outcome: Number of Participants With Disease Progression or Recurrence of GCTB
Description: Disease progression or recurrence is defined as the best post-baseline response of progressive disease (PD) without any post-baseline complete response (CR) /partial response (PR) /stable disease (SD) or a post-baseline response of PD following a post-baseline CR/PR/SD. PD is defined as the response of progressive disease, locally recurrent disease or distant recurrence. CR is defined as no evidence of disease following surgical resection while on study 20062004. PR is defined as no new lesion or disease progression while enrolled in study 20062004. SD is defined as local disease progression/recurrence or distant metastatic disease while on study 20062004.
Time Frame: Up to approximately 5 years
Population: FAS included all enrolled participants (from study 20062004) who provided informed consent and had a non-missing enrolment date in this study. The number of participants analyzed is inclusive of participants with available data.
Measure: Number; unit: Count of Participants
Arm/Group | Exposed to IP | Not Exposed to IP
Number analyzed (Participants) | 50 | 33
Count of Participants | 5 | 3

4. Secondary Outcome: Number of Participants Receiving GCTB Interventions
Description: GCTB interventions include: surgery, chemotherapy, embolization, interferon, and radiotherapy.
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Measure: Number; unit: Count of Participants
Arm/Group | Exposed to IP | Not Exposed to IP
Number analyzed (Participants) | 51 | 34
Count of Participants
  Surgery for GCTB | 1 | 3
  Chemotherapy or Other Therapeutic Agents | 0 | 2
  Embolization | 0 | 0
  Interferon | 0 | 0
  Radiotherapy | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Approximately 5 years
Description: FAS included all enrolled participants (from study 20062004) who provided informed consent and had a non-missing enrolment date in this study.
Groups:
- Exposed to IP: Subjects treated with study IP
- Not Exposed to IP: Subjects not treated with study IP
Arm/Group | Exposed to IP | Not Exposed to IP
All-Cause Mortality (participants affected / at risk) | 0/51 | 2/34
Serious Adverse Events (participants affected / at risk) | 8/51 | 0/34
Other Adverse Events (participants affected / at risk) | 37/51 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exposed to IP (N=51) | Not Exposed to IP (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Medical device site infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exposed to IP (N=51) | Not Exposed to IP (N=34)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Toothache (Gastrointestinal disorders) | 8 | 0
Pyrexia (General disorders) | 3 | 0
COVID-19 (Infections and infestations) | 7 | 0
Gingivitis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 0
Headache (Nervous system disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03301857/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03301857/SAP_001.pdf